CLINICAL TRIAL: NCT03354208
Title: Verification of Biomarkers to Examine Neonatal Asphyxia Induced Hypoxic-ischemic Encephalopathy. A Prospective Multicenter Observational Study for Development of a Diagnostic Test
Brief Title: Asphyxia Associated Metabolite Biomarker Investigation (AAMBI)
Acronym: AAMBI
Status: Completed | Type: Observational
Sponsor: Life Science Inkubator (Other)
Collaborators: Cukurova University (Other); University Children's Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: AAMBI I
Record Dates: First submitted 2017-09-22; First posted 2017-11-27 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Asphyxia Neonatorum
Keywords: biomarkers
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: patients with hypoxic-ischemic encephalopathy (HIE) receiving hypothermia therapy
  Interventions: Other: blood sampling
- Group 2: patients with suspected HIE, non-confirmed
  Interventions: Other: blood sampling
- Group 3: healthy, retrospectively classified as such
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — small volume blood sampling, according to local laws, is not categorized as intervention (observational study)

SUMMARY:
Verification of biomarkers in a human population for their ability to diagnose the severity of neonatal asphyxia. These biomarkers linked to asphyxia have been identified in animal studies.

DETAILED DESCRIPTION:
The aim of the study is to verify the application of combinations of several laboratory parameters in early postnatal blood samples, for identification of infants, who will suffer from early abnormal neonatal neurological outcome, in a population at risk.

The population at risk is defined as term and late preterm (>36 weeks of gestation) human infants following perinatal hypoxia-ischemia with or without postnatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

Group 1: inclusion criteria fulfilled for hypothermia treatment Group 2: Infants with suspected perinatal brain injury due to one of the followings

* Perinatal hypoxia-ischemia (defined as a perinatal acidosis indicated by a pH≤7.10 or a base excess ≤-12mmol/l in umbilical cord blood or early postnatal blood collected at <90min of age (outborn patients)
* 5min APGAR-score ≤ 5
* Need for resuscitation after birth for >1 min. after birth, positive pressure respiratory support with face mask or endotracheal tube, or cardiac compressions Group 3: UApH >7,25, and adaptation disorder of the newborn and need of postnatal clinical surveillance

Exclusion Criteria:

gestational age < 36 weeks

* age at time of screening >2,5h
* congenital malformation
* missing or invalid informed parental consent
* unsuccessful resuscitation
* infant considered not-viable
* decision for palliative care only

Ages: 0 Hours to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants at risk for perinatal hypoxic-ischemic brain injury
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
abnormal short-term outcome (NE) | 14 days for clinical diagnosis
  All patients are classified as abnormal short-term outcome (neonatal encephalopathy, NE) or normal short term outcome (no encephalopathy) by using clinical data, particularly Thompson score. For Group 1 and group 2 patients outcome classification will be additionally confirmed by using cranial ultrasound or MRI (including severe ischemia based on DWI or thalamic or cerebellar bleeding or arterial infarction or IVH>2° according to Papile, thalamic ischemia or severe cerebral edema) or seizure activity or burst suppression on aEEG or persistingly abnormal aEEG background pattern after complete rewarming.
  Bloodplasma samples will be analysed by a metabolomics approach using the p180-kit (Biocrates, Innsbruck, Austria). Metabolite concentrations or combinations thereof will be compared to the outcome described above in order to identify the most suitable metabolites to be used for early detection of NE in newborn infants.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Meyer, Study Director — Life Science Inkubator Betriebs GmbH & Co. KG
Locations (4):
- Turkey (Türkiye) (4):
  - Cukurova University, Adana
  - University of Firat, Elâzığ
  - Özel Güngören Hastanesi, Istanbul
  - Mersin University School of Medicine, Mersin

IPD SHARING:
Plan to Share IPD: No